CLINICAL TRIAL: NCT02121314
Title: The Influence of Fasting and Food on the Pharmacokinetics of Isoniazid, Rifampicin, Pyrazinamide, and Ethambutol in Newly Diagnosed TB Patients
Brief Title: HRZE Fasted/Fed in Newly Diagnosed TB
Acronym: FASTFOOD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: University of Groningen (Other); Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Tjip van der Werf, Professor, Infectious Diseases & Tuberculosis, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UGM-RuG-UMCG-TB-001
Record Dates: First submitted 2014-01-25; First posted 2014-04-23 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Tuberculosis
Keywords: TB; bioavailability; HRZE; fasting; fed
MeSH Terms: conditions — Tuberculosis; Fasting; Lecithin Cholesterol Acyltransferase Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fasting-Fed (Active Comparator): blood sampling on 3 consecutive days; by randomization, drug treatment as follows: day 1, HRZE as iv therapy; on day 2, HRZE as oral therapy in fasting condition (2 hours before meals); and on day 3 HRZE as oral therapy in fed condition (after meals).
  Interventions: Drug: intravenous administration of 1st line TB drugs, day 1
- Fed-Fasting (Active Comparator): blood sampling on 3 consecutive days; by randomization, drug treatment as follows: day 1, HRZE therapy as iv therapy; day 2, HRZE as oral therapy in fed condition, and on day 3, HRZE as oral therapy in fasting condition
  Interventions: Drug: intravenous administration of 1st line TB drugs, day 1

INTERVENTIONS:
Drug: intravenous administration of 1st line TB drugs, day 1 — TB drugs IV on day 1 for calculation of bioavailability while fasting or fed

SUMMARY:
WHO recommends to take TB drugs while fasting: if TB drugs are taken with food, perhaps drug concentrations are too low; on the other hand: if this is not tolerated, drugs could also be taken with food.

Do lower drug concentrations - with improved adherence to therapy - outweigh the disadvantage of lower drug blood concentrations over time? How exactly do the drug concentrations over time (pharmacokinetics) compare between fasting and fed conditions, especially in the early stage of TB treatment when patients are relatively sick, and relatively poorly tolerate TB drugs?

DETAILED DESCRIPTION:
To evaluate the influence of concomitant food ingestion on the pharmacokinetics of HRZE in newly diagnosed TB patients To evaluate the influence of early disease on the PK parameters of HRZE in TB patients To compare the pharmacokinetics of HRZE in the early stage of disease with the pharmacokinetics of HRZE in more stable condition in newly diagnosed TB patients To evaluate adverse events of HRZE in TB patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with TB who are starting with HRZE therapy
* Age > 18 years old
* Written informed consent

Exclusion Criteria:

* Use of antacids, which cannot be discontinued for study days
* Active, unstable hepatic disease (with jaundice, HRZ)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics | 3 days - week 1 and week 8
  pharmacokinetics (AUC0-8, Cmax, and Tmax); comparison between TB patients who take HRZE concomitant with food and TB patients who take HRZE concomitant without food, weeks 1 and 8 of treatment
pharmacokinetics (AUC0-8, Cmax, and Tmax) of HRZE | 11 time points, 3 consecutive days - wk 1 & 8
  PK curves from venous blood specimens sampled from indwelling venous catheter

SECONDARY OUTCOMES:
To evaluate adverse events of HRZE, week 1 and 8 - while taking food or not | week 1 - week 8
  tolerance - acceptance; vomiting, refusal

OTHER OUTCOMES:
confounding factors for primary and secondary outcomes | weeks 1 and 8
  Parameters which may influence the pharmacokinetics of HRZE will be measured at start and end of the study.
  * BMI, i.e. body weight and length
  * age
  * gender
  * ethnicity
  * co-morbidity, for instance HIV/AIDS, diabetes (only at start)
  * co-medication: especially HIV medication, prednisolone (may lower INH concentration), antacids (may lower absorption of HRE concentration)
  * chemistry: liver function, renal function, hemoglobulin, albumin, bilirubin
  * pharmacogenetics

CONTACTS AND LOCATIONS:
Locations (1):
- Sardjito Central Hospital, Yogyakarta, Indonesia

REFERENCES:
- [Derived] Saktiawati AMI, Harkema M, Setyawan A, Subronto YW, Sumardi, Stienstra Y, Aarnoutse RE, Magis-Escurra C, Kosterink JGW, van der Werf TS, Alffenaar JC, Sturkenboom MGG. Optimal Sampling Strategies for Therapeutic Drug Monitoring of First-Line Tuberculosis Drugs in Patients with Tuberculosis. Clin Pharmacokinet. 2019 Nov;58(11):1445-1454. doi: 10.1007/s40262-019-00763-3. PMID 30997650
- [Derived] Saktiawati AM, Sturkenboom MG, Stienstra Y, Subronto YW, Sumardi, Kosterink JG, van der Werf TS, Alffenaar JW. Impact of food on the pharmacokinetics of first-line anti-TB drugs in treatment-naive TB patients: a randomized cross-over trial. J Antimicrob Chemother. 2016 Mar;71(3):703-10. doi: 10.1093/jac/dkv394. Epub 2015 Dec 11. PMID 26661397